CLINICAL TRIAL: NCT06662851
Title: Usefulness of Ultrasound-derived Fat Fraction for Quantification of Hepatic Steatosis in Patients Suspected of MASLD: a Prospective Study
Brief Title: Usefulness of Ultrasound-derived Fat Fraction for Quantification of Hepatic Steatosis in Patients Suspected of MASLD
Status: Active, not recruiting | Type: Observational
Sponsor: So Yeon Kim (Other)
Responsible Party: Sponsor-Investigator, So Yeon Kim, MD, PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: ASANMC_UDFF
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease
Keywords: MASLD; Ultrasound; Steatosis; Liver Diseases; Fibrosis
MeSH Terms: conditions — Fatty Liver; Liver Diseases; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pathological degree of hepatic steatosis and fibrosis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: UDFF — Ultrasound-Derived Fat Fraction (UDFF) is a quantitative ultrasound technique used to assess hepatic steatosis by measuring the amount of fat in the liver tissue. UDFF estimates fat content using specific ultrasound parameters, namely the attenuation coefficient (AC) and backscatter coefficient (BSC). The AC measures the rate at which ultrasound waves weaken as they pass through the liver, which correlates with fat content, while the BSC quantifies the amount of reflected ultrasound signal, providing additional insights into liver tissue characteristics.

SUMMARY:
This study aims to evaluate the diagnostic utility of ultrasound-derived fat fraction (UDFF) in assessing hepatic steatosis in patients with suspected metabolic dysfunction-associated steatotic liver disease (MASLD). Using a prospective, cross-sectional design, the study will compare UDFF results with established diagnostic methods, including liver biopsy, MRI proton density fat fraction (PDFF), and controlled attenuation parameters (CAP) measurements. The ultimate goal is to determine if UDFF can serve as a non-invasive alternative to liver biopsy for diagnosing and staging hepatic steatosis, potentially reducing the need for invasive procedures in MASLD management.

DETAILED DESCRIPTION:
This prospective observational study, conducted at a single tertiary institution, will investigate the efficacy of ultrasound-derived fat fraction (UDFF) and point shear wave elastography (p-SWE) as non-invasive methods for quantifying liver fat content and fibrosis in patients scheduled for liver biopsy or surgery. The study will enroll 150 participants, suspected of MASLD and who are candidates for liver biopsy or resection.

The study will utilize Siemens ultrasound equipment to measure the UDFF using attenuation coefficient (AC) and backscatter coefficient (BSC) values for liver fat quantification. Additionally, TE parameters, such as controlled attenuation parameter (CAP) and liver stiffness measurement (LSM), will be recorded for comparison. The primary outcomes will assess UDFF's diagnostic accuracy against liver biopsy and MRI-PDFF. Secondary outcomes will include assessment of intra- and inter-observer variability, and correlations with patients' clinical data, such as BMI, liver fibrosis stages and liver function tests.

Expected benefits include validating UDFF as a reliable, non-invasive alternative for liver fat assessment, potentially reducing the need for invasive biopsies in managing liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 and younger than 80 years
* Patients suspected of MASLD
* Patients who are planned to undergo either liver biopsy or surgery
* Patients willing to provide written informed consent.

Exclusion Criteria:

* Patients with a large tumor in Rt. hemiliver causing difficulty in performing UDFF measurement
* Patients with previous liver surgery or transplantation
* Patients with insufficient pathologic specimen for analysis of steatosis and fibrosis grade.
* Any other condition which, in the opinion of the investigator, would make the patient unsuitable for enrollment or could interfere with completing the study.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected of MASLD, who are scheduled for pathologic exam such as liver biopsy or surgery
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Correlation and agreement between UDFF and PDFF | During procedure
  Spearman rank correlation coefficient Intraclass correlation coefficient (ICC) with a 2-way random effects model for absolute agreement Bland-Altman plots
Diagnostic performance of UDFF for detecting and grading steatosis based on PDFF and histologic reference | During procedure
  AUROC analysis

SECONDARY OUTCOMES:
Intra-observer and inter-observer agreement | During procedure
  Intraclass correlation coefficient
UDFF performance in different fibrosis stages | During procedure
  Subgroup analysis according to different fibrosis stages

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No